CLINICAL TRIAL: NCT01245335
Title: Pivotal Study of the Safety and Effectiveness of Autologous Bone Marrow Aspirate Concentrate (BMAC) for the Treatment of Critical Limb Ischemia Due to Peripheral Arterial Disease
Brief Title: Bone Marrow Aspirate Concentrate (BMAC) for Treatment of Critical Limb Ischemia (CLI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLI-2011-1
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Critical Limb Ischemia
Keywords: CLI; Critical Limb Ischemia; PAOD; Peripheral Arterial Disease; Stem Cells; Limb amputation; Leg ulcers
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease; Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BMAC Treatment (Active Comparator): Intervention- Injection of 40 ml of autologous bone marrow concentrate (BMAC injection) prepared with the SmartPReP2 BMAC System
  Interventions: Device: BMAC injection
- Placebo Injection (Placebo Comparator): Injection of placebo (diluted peripheral blood) into ischemic tissue of the lower extremity
  Interventions: Device: Placebo injection

INTERVENTIONS:
Device: BMAC injection — Injection of 40 ml of autologous bone marrow aspirate concentrate (BMAC injection) prepared with the SmartPReP2 BMAC System
  Arms: BMAC Treatment
Device: Placebo injection — Injection of placebo into ischemic tissue of the lower extremity
  Arms: Placebo Injection

SUMMARY:
Critical Limb Ischemia prevents the legs and feet from receiving oxygen and nutrients needed for proper function. This severe lack of blood flow can lead to painful legs while walking or at rest and can result in foot sores, ulcers, gangrene, and even amputation. The purpose of this study is to determine if injections of concentrated bone marrow into damaged tissues will result in improved blood flow. If successful, this treatment could improve blood flow to the lower limb, reduce pain, and reduce the frequency of limb amputations.

DETAILED DESCRIPTION:
Bone marrow aspirate is collected and processed by centrifugation to remove red blood cells. The resulting concentrate of cells is injected into ischemic tissues of the lower limb. The purpose of this study is to determine if injections of concentrated bone marrow nucleated cells into ischemic tissues will result in vasculogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Peripheral Arterial Occlusive Disease (PAOD) with clinical Rutherford Category 5 disease, as defined in the reporting standards adopted by the Society of Vascular Surgeons(table 1); Minor Tissue loss-focal gangrene with diffuse pedal ischemia
* Patient meets at least one of the following diagnostic criteria in the study limb:

  * Ankle artery occlusion pressure absolute ≤60 mmHg or ABI ≤0.6
  * Toe artery occlusive pressure < 50mm Hg or TBI ≤0.6
* There is no reasonable open surgical or endovascular revascularization option as determined by the treating vascular specialist. Factors that may contribute to the determination of inoperability may include:

  * Anatomical considerations
* No outflow targets
* No appropriate conduit (i.e. vein for bypass)
* Long segment occlusions or calcified lesions that predict poor outcome with endovascular approaches.

  * High risk medical conditions i.e. Unstable cardiac disease.
  * History of prior failed revascularization attempts
* The Patient's case was reviewed at the treating institution's Multidisciplinary Vascular Conference where the patient's status as a poor candidate for conventional therapies was confirmed.
* Age ≥18 years and ability to understand the planned treatment
* Subject has read and signed the IRB approved Informed Consent form
* Patients for whom the following medication(s) is prescribed must have a one month stable baseline therapy prior to enrollment: Plavix/asprin therapy, anticoagulation therapy, cholesterol lowering agent, and or blood pressure medication. If any of these medications are not prescribed notation of the reason for omission is to be provided.
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, Creatinine ≤ 2.5 mg / dL, INR ≤ 1.6 unless on Coumadin, or PTT <1.5 x control (to avoid bleeding complications) Patients on Coumadin will be corrected prior to the procedure and must have an INR<1.6 at the time of randomization/surgery.

Exclusion Criteria:

* Life expectancy <6 months due to concomitant illnesses
* History of bone marrow diseases (especially NHL, MDS) that prohibit transplantation
* Terminal renal failure with existing dependence on dialysis or serum creatinine >2.5 mg/dL
* Known active malignancy or results outside of normal limits from the following tests: PAP, Chest X-ray, PSA, Mammogram, Hemocult unless follow-up studies reveal patient to be cancer free.
* Poorly controlled diabetes mellitus (HgbA1C>10%)
* Medical risk that precludes anesthesia (conscious sedation), or ASA Class 5
* Life-threatening complications of the ischemia necessitating immediate amputation
* Uncorrected occlusion of the common or external iliac artery on index side
* Absence of any pulsatile Doppler flow below the ankle.
* Extensive necrosis of the index limb or other conditions that make amputation inevitable (Rutherford Category 6).
* Ulceration with exposed bone proximal to the distal metatarsal heads (ie. heel or mid foot)
* Active clinical infection or infection being treated by antibiotics within one week of enrollment
* Treatment with immunosuppressant drugs (including Prednisone > 5 mg per day).
* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method.
* Underwent a major open cardiovascular surgical procedure (carotid endarterectomy, arterial aneurysm or bypass surgery, or coronary artery bypass surgery) or a myocardial infarction within the 3 months prior to randomization
* Underwent a successful or partially successful endovascular intervention for peripheral arterial occlusive disease. (ie. Aorta, iliac, femoral, popliteal, or tibial artery angioplasty, stenting, or atherectomy) within the prior 3 months.
* Endovascular coronary intervention (ie. Angioplasty, atherectomy, stenting) within 1 month prior to randomization.
* Underwent a failed attempt for endovascular revascularization during the prior 1 month. For the purpose of this exclusion criteria an endovascular procedure is considered a failure if:

  1. The procedure is diagnostic only with no intervention performed, (for example in the case where wire crossing can not be obtained).
  2. The treated artery recoils, thromboses, or dissects resulting in occlusion of the treated arterial segment, documented by intraoperative imaging. Note that endovascular procedures with suboptimal results but not meeting criteria 1 or 2 above may qualify for inclusion after 3 months as in #16 above.
* Cerebrovascular accident within 6 months prior to randomization.
* Treatment with topical growth factors or hyperbaric oxygen (HBO) within 30 days, or systemic growth factor treatment within 6 months of enrollment.
* Known hypersensitivity to heparin; or history of heparin-induced thrombocytopenia (HIT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Amputation Free Survival | Six Months
  Survival without a major (above the ankle) amputation

SECONDARY OUTCOMES:
Change In Rutherford Classification | Six Months
  Change in the subjects clinical status as measured by Rutherford Classification
Change in Pain | Six Months
  Change in Subjects perception of pain as measured on a 100 mm visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark Iafrati, MD, Principal Investigator — Tufts Medical Ctr
Locations (34):
- United States (34):
  - University of Alabama, Birmingham, Alabama
  - Medical Center of South Arkansas, El Dorado, Arkansas
  - USC Keck School of Medicine, Los Angeles, California
  - Florida Hospital - Vascular Institute of Central Florida, Orlando, Florida
  - Coastal Vascular & Interventional, Pensacola, Florida
  - USF / Tampa General, Tampa, Florida
  - University of Illinois-Chicago, Chicago, Illinois
  - Cadence Health, Central DuPage Hospital, Winfield, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Ctr, Portland, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Kansas City Vascular, Kansas City, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Ctr, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - North Shore-Long Island Jewish, Lake Success, New York
  - St. Luke's Roosevelt, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Regional Infectious Disease and Infusion Ctr, Lima, Ohio
  - University of Oklahoma, Tulsa, Oklahoma
  - Oregon Health Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Roper St Francis Medical Center, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - University of Tennessee, Knoxville, Tennessee
  - Baylor Medical Ctr, Dallas, Texas
  - University of Texas - Houston Medical School, Houston, Texas
  - Peace Health Southwest Medical Center, Vancouver, Washington
  - Charleston Area Medical Center Institute, Charleston, West Virginia